CLINICAL TRIAL: NCT02070237
Title: Comparing Anti-XA Levels in Post-Cesarean Patients With BMI >35 Undergoing Enoxaparin Thromboprophylaxis With Weight Based Dosing Twice Daily Versus Fixed Dose 40 Milligrams Daily
Brief Title: Comparing Anti-XA Levels in Post-Cesarean Patients Undergoing Enoxaparin Thromboprophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 159-12
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-01

CONDITIONS: Obesity; Obesity, Morbid; Pregnancy; Complications; Cesarean Section; Venous Thromboembolism; Postpartum Deep Phlebothrombosis; Pulmonary Embolism
Keywords: Obesity; Obesity, Morbid; Pregnancy; Cesarean; Venous thromboembolism; Deep venous thrombosis; Pulmonary embolism
MeSH Terms: conditions — Obesity; Obesity, Morbid; Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin Once Daily (Active Comparator): This arm will have patients randomized to receive 40 mg sub-cutaneous injection of Lovenox (enoxaparin) once daily.
  Interventions: Drug: Enoxaparin
- Enoxaparin Twice Daily (Active Comparator): This arm will have patients randomized to receive weight based (0.5 mg/kg) sub-cutaneous injection of Lovenox (enoxaparin) twice daily.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin will be given in either once daily or twice daily doses. One arm will receive 40 mg enoxaparin subcutaneous injection daily. The other arm will receive 0.5 mg/kg dosed subcutaneously twice daily. This medication will be started 8-12 hours after cesarean section and will be continued while the patient is admitted. It will be stopped at the time of discharge.
  Other Names: Lovenox

SUMMARY:
Pregnant and recently postpartum women are at significantly higher risk of developing a blood clot in their arms or legs known as a deep venous thrombosis (DVT) and/or a blood clot in their lungs known as a pulmonary embolism (PE) compared to their non pregnant counterparts. It is estimated that this risk increases anywhere from 4 to 50 times higher in pregnant versus non-pregnant women and further increases almost 11 fold in the post partum period. This risk is almost doubled when the patient undergoes cesarean delivery. In 2011, the American College of Obstetricians and Gynecologists (ACOG) issued updated guidelines stating that for patients undergoing cesarean delivery with additional risk factors for clot or thromboembolism, protective (prophylactic) treatment with low molecular weight heparin (LMWH) a type of blood thinner should be considered. However, no specific guidelines about which risk factors should be considered, or what medication doses should be used were provided. The American College of Chest Physicians (ACCP) Evidence-Based Clinical Practice Guidelines published in 2012 delineated who should be given prophylaxis based on various risk factors, however acknowledged that the recommendations were based on weak quality evidence.

ACOG endorses either once or twice a day dosing for high risk patients after delivery and states that adjustments for obese women should be made on a case by case basis. However, there are limited studies on the dosing of LMWH in specific subpopulations including post operative patients, pregnant patients and obese patients. All of these studies have urged further investigation of the correct dosing for these high risk subjects due to changes associated with pregnancy and the level of medication in the blood that may put these patients at higher risk of venous thromboembolism. Many previous studies have shown that women in these high risk categories do not achieve protective levels of the medication measured with a laboratory test; anti Xa level. The investigators hypothesize that due to their dual risk, obese post-operative recently pregnant women may not be adequately protected with the daily fixed dose and might need more frequent dosing to protect them.

The objective of this study is to assess what proportion of women achieve the desired anti Xa level with the fixed daily dose versus twice daily weight based dosing (0.5 mg/kg).

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized controlled study to compare the proportion of patients that achieve the desired effect of LMWH (enoxaparin) thromboprophylaxis as measured by peak anti Xa level with weight based twice daily dosing versus standard fixed daily dosing. The investigators hypothesize that when enoxaparin is dosed by maternal weight and administered twice daily, the anti-factor Xa level would more frequently achieve prophylactic levels when compared to taking a fixed 40 mg of the drug daily.

Subjects will be women with a BMI > 35 who have undergone a cesarean delivery and who will receive thromboprophylaxis with enoxaparin (Lovenox) at the judgment of their physician.

Women who are eligible and consent to participate in the study will be randomized in a 1:1 ratio to one of the following groups:

Group 1 will receive the weight based dosing (0.5mg/kg BID) enoxaparin (Lovenox®; Aventis Pharmaceuticals) regimen Group 2 will received the fixed dose (40mg daily) enoxaparin (Lovenox®; Aventis Pharmaceuticals) regimen.

Treatment will begin between 8 and 12 hours post operatively and this regimen will continue until discharge from the hospital, usually on the third or fourth day after surgery. A single peak anti Xa level will be drawn 3.5-4 hours after the third dose of medication. The results of the anti Xa level will only be for research purposes and will not guide clinical management.

The primary outcome for this study is to assess the peak anti-factor Xa level in the blood, and whether or not the subject achieved the desired prophylactic level when receiving fixed dose of enoxaparin compared with weight based dosing.

ELIGIBILITY:
Inclusion Criteria:

* Women with a body mass index >35 who have undergone cesarean delivery in the last 12 hours who will receive thromboprophylaxis with enoxaparin
* Subjects who consent to the study.

Exclusion Criteria:

* Women with a previous history of deep venous thrombosis or pulmonary embolism
* Women who are currently receiving another form of low molecular weight heparin or unfractionated heparin.
* Women who are receiving other concomitant anticoagulant medications, such as warfarin, lepirudin, or argatroban.
* Subjects who are unable or unwilling to give informed consent.
* Women who, in the judgment of the investigators, would not be in the best interest of the patient to participate in the study.
* Allergy to enoxaparin.
* Women with renal impairment
* Women with contraindications to Lovenox treatment such as women with active bleeding or thrombocytopenia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNulty, MD, Principal Investigator — Memorial Care Health System; Megan L Stephenson, MD, Principal Investigator — Memorial Health Care System; University of California Irvine
Locations (1):
- Long Beach Memorial Care Center for Women at Miller Children's Hospital Long Beach and Long Beach Memorial Hospital, Long Beach, California, United States

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Stephenson ML, Serra AE, Neeper JM, Caballero DC, McNulty J. A randomized controlled trial of differing doses of postcesarean enoxaparin thromboprophylaxis in obese women. J Perinatol. 2016 Feb;36(2):95-9. doi: 10.1038/jp.2015.130. Epub 2015 Dec 10. PMID 26658126

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enoxaparin Once Daily | Enoxaparin Twice Daily
Started | 45 | 45
Completed | 42 | 42
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin Once Daily | Enoxaparin Twice Daily | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.6) | 30 (5.4) | 32 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Anti Xa Level
Description: Our primary outcome will be to assess the Anti Xa level drawn 3.5-4 hours after the third dose of Lovenox (enoxaparin) to assess if this is in the prophylactic range.
Time Frame: 3.5-4 hours after the third dose of Lovenox (enoxaparin)
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Enoxaparin Once Daily | Enoxaparin Twice Daily
Number analyzed (Participants) | 42 | 42
IU/mL | 0.14 [0.12 to 0.16] | 0.30 [0.27 to 0.31]

2. Secondary Outcome: Supraprophylactic Range Anti Xa Level
Description: We will assess if any of the subjects has an Anti Xa level that is in the supraprophylactic range (treatment range).
Time Frame: 3.5-4 hours after the third dose of Lovenox (enoxaparin)
Measure: Number; unit: participants
Arm/Group | Enoxaparin Once Daily | Enoxaparin Twice Daily
Number analyzed (Participants) | 42 | 42
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Enoxaparin Once Daily | Enoxaparin Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No